CLINICAL TRIAL: NCT02140554
Title: A Phase 1/2 Study Evaluating Gene Therapy by Transplantation of Autologous CD34+ Stem Cells Transduced Ex Vivo With the LentiGlobin BB305 Lentiviral Vector in Subjects With Severe Sickle Cell Disease
Brief Title: A Study Evaluating the Safety and Efficacy of Lovo-cel in Severe Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGB-206
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — lyfgenia; Excipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Participants who had rescue cells that were collected by bone marrow harvest method and had received treatment with lovo-cel which consists of autologous CD34+ hematopoietic stem cells (HSCs) and progenitor stem cells (PSCs) (collectively referred to as hematopoietic stem and progenitor cells or HSPCs) collected from participants with sickle cell disease (SCD) by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene (the original drug product manufacturing process for this study).
  Interventions: Genetic: lovo-cel
- Group B (Experimental): Group B1 participant had rescue cells and drug product cells that were collected by bone marrow harvest method and drug product was manufactured with autologous CD34+ HSPCs collected by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene. This participant's drug product was produced in 2 lots each using two different manufacturing processes (the original drug product manufacturing process and a refined drug product manufacturing process).
  Group B2 Plerixafor mobilization and apheresis were used for collection of rescue cells and exploratory manufacturing development. A single Group B2 participant received treatment of lovo-cel manufactured with autologous CD34+ HSPCs collected by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene (using only the refined drug product manufacturing process).
  Note: Groups B1 and B2 are combined as "Group B" for results reporting purposes.
  Interventions: Genetic: lovo-cel
- Group C (Experimental): Plerixafor mobilization and apheresis were used for collection of rescue cells, and drug product. Participants received treatment of lovo-cel manufactured with autologous CD34+ HSPCs collected by plerixafor mobilization and apheresis transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene using a further refined manufacturing process similar to commercial manufacturing.
  Interventions: Genetic: lovo-cel

INTERVENTIONS:
Genetic: lovo-cel — lovo-cel is administered by IV infusion following myeloablative conditioning with busulfan.
  Other Names: lovotibeglogene autotemcel; bb1111; LentiGlobin BB305 Drug Product for SCD; autologous CD34+ cell-enriched population with SCD that contains HSCs and PSCs transduced with BB305 lentiviral vector encoding the βA-T87Q-globin gene, suspended in cryopreservation solution.

SUMMARY:
This is a non-randomized, open label, multi-site, single dose, Phase 1/2 study in approximately 50 adults and adolescents with severe SCD. The study will evaluate hematopoietic stem cell and progenitor stem cell (collectively referred to as hematopoietic stem and progenitor cells or HSPCs) transplantation using lovo-cel.

DETAILED DESCRIPTION:
Subject participation for this study will be 2 years post-transplant. Subjects who enroll in this study will be asked to participate in a subsequent long-term follow up study that will monitor the safety and efficacy of the treatment they receive for an additional 13 years for a total of 15 years post-drug product infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥12 and ≤50 of age at time of consent.
2. Diagnosis of sickle cell disease (SCD), with either βS/βS or βS/β0 or βS/β+ genotype.
3. Have severe SCD. i.e., in the setting of appropriate supportive care measures for SCD (e.g., pain management plan), have experienced at least 4 severe VOEs in the 24 months prior to informed consent.

   For the purposes of this study, a severe VOE is defined as an event with no medically determined cause other than a vaso-occlusion, requiring a ≥ 24-hour hospital or Emergency Room (ER) observation unit visit or at least 2 visits to a day unit or ER over 72 hours with both visits requiring intravenous treatment. Exception: priapism does not require hospital admission but does require a medical facility visit; 4 priapism episodes that require a visit to a medical facility (without inpatient admission) are sufficient to meet criterion.

   Severe VOEs include:
   1. an episode of acute pain with no medically determined cause other than a VOE
   2. Acute chest syndrome (ACS), defined by an acute event with pneumonia-like symptoms (e.g., chest pain, fever [> 38.5°C], tachypnea, wheezing or cough, or findings upon lung auscultation) and the presence of a new pulmonary infiltrate consistent with ACS and requiring oxygen treatment and/or blood transfusion.
   3. Acute hepatic sequestration, defined by a sudden increase in liver size associated with pain in the right upper quadrant, abnormal results of liver-function test not due to biliary tract disease, and reduction in Hb concentration by at least 2 g/dL below the baseline value
   4. Acute splenic sequestration, defined as sudden enlargement of the spleen and reduction in Hb concentration by at least 2 g/dL below the baseline value.
   5. Acute priapism: defined as a sustained, unwanted painful erection lasting more than 2 hours and requiring care at a medical facility (with or without hospitalization)
4. Karnofsky performance status of ≥ 60 (≥16 years of age) or a Lansky performance status of ≥60 (<16 years of age).
5. Have either experienced hydroxyurea (HU) failure at any point in the past or must have intolerance to HU (defined as patient being unable to continue to take HU per PI judgement).
6. Have been treated and followed for at least the past 24 months prior to Informed Consent in medical center(s) that maintained detailed records on SCD history.

Exclusion Criteria:

1. Positive for presence of human immunodeficiency virus type 1 or 2 (HIV-1 and HIV-2), hepatitis B virus (HBV), or hepatitis C (HCV).
2. Clinically significant and active bacterial, viral, fungal, or parasitic infection.
3. Inadequate bone marrow function, as defined by an absolute neutrophil count of < 1000/µL (< 500/µL for subjects on HU treatment) or a platelet count < 100,000/µL.
4. Any history of severe cerebral vasculopathy: defined by overt or hemorrhagic stroke; abnormal transcranial Doppler [≥200 cm/sec] needing chronic transfusion; or occlusion or stenosis in the polygon of Willis; or presence of Moyamoya disease. Subjects with radiologic evidence of silent infarction in the absence of any of the above criteria would still be eligible
5. Baseline oxygen saturation < 90% without supplemental oxygen (excluding periods of SCD crisis, severe anemia or infection).
6. Baseline carbon monoxide diffusing capacity (DLCO) < 50% (corrected for Hb) in the absence of infection. If DLco cannot be assessed due to age or cognition-related restrictions, there must be a normal respiratory exam, chest radiograph without pulmonary infiltrates, and oxygen saturation by pulse oximetry ≥ 90% on room air.
7. Baseline left ventricular ejection fraction (LVEF) < 45% measured by cardiac echography.
8. Clinically significant pulmonary hypertension at baseline, as defined by the requirement for ongoing pharmacologic treatment or the consistent or intermittent use of supplemental home oxygen.
9. Baseline estimated glomerular filtration rate (eGFR) < 70 mL/min/1.73 m2, as determined using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (see http://www.kidney.org/professionals/kdoqi/gfr_calculator.cfm).
10. Advanced liver disease, defined as:

    1. Persistent aspartate transaminase, alanine transaminase, or direct bilirubin value >3× the upper limit of normal (ULN), or
    2. Baseline prothrombin time or partial thromboplastin time >1.5× ULN, suspected of arising from liver disease, or
    3. Magnetic Resonance Imaging (MRI) of the liver demonstrating clear evidence of cirrhosis, or
    4. MRI findings suggestive of active hepatitis, significant fibrosis, inconclusive evidence of cirrhosis, or liver iron concentration ≥15 mg/g require follow-up liver biopsy in subjects ≥18 years of age. In subjects <18 years of age, these MRI findings are exclusionary, unless in the opinion of the Investigator, a liver biopsy could provide additional data to confirm eligibility and would be safe to perform. If a liver biopsy is performed based on MRI findings, any evidence of cirrhosis, bridging fibrosis, or significant active hepatitis will be exclusionary.
11. For subjects who have history of iron overload or serum ferritin levels > 1000 ng/mL, a cardiac MRI is required. Cardiac T2* < 10 ms results in exclusion.
12. Contraindication to anesthesia.
13. Any contraindications to the use of plerixafor during the mobilization of hematopoietic stem cells and any contraindications to the use of busulfan and any other medicinal products required during the myeloablative conditioning, including hypersensitivity to the active substances or to any of the excipients.
14. Any prior or current malignancy or immunodeficiency disorder, except previously treated, non-life threatening, cured tumors such as squamous cell carcinoma of the skin.
15. Prior receipt of an allogeneic transplant.
16. Immediate family member with a known or suspected Familial Cancer Syndrome.
17. Diagnosis of significant psychiatric disorder of the subject that, in the Investigator's judgment, could seriously impede the ability to participate in the study.
18. Pregnancy or breastfeeding in a postpartum female or absence of adequate contraception for fertile subjects.
19. Participation in another clinical study with an investigational drug within 30 days of Screening.
20. Prior receipt of gene therapy.
21. An assessment by the Investigator that the subject or parents/caregivers (as required) will not be able to comply with the study procedures outlined in the study protocol.
22. Patients needing therapeutic anticoagulation treatment during the period of conditioning through platelet engraftment (patients on prophylactic doses of anticoagulants not excluded per this criteria).
23. Unable to receive Red Blood Cell (RBC) transfusion.
24. Any other condition that would render the subject ineligible for hematopoietic stem cell transplant (HSCT), as determined by the attending transplant physician.
25. Applicable to subjects < 18 years of age only: Availability of a willing, matched HLA-identical sibling hematopoietic cell donor.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjulika Chawla, MD, FAAP, Study Director — bluebird bio, Inc.
Locations (11):
- United States (11):
  - Birmingham, Alabama
  - Oakland, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Bethesda, Maryland
  - Hackensack, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency. Appropriately de-identified patient-level datasets and supporting documents may be shared (if contractually or otherwise legally permitted) following study completion and and once all applicable regulatory submissions based on this study have been performed. Sharing of individual patient data will be done according to criteria established by bluebird bio and/or industry best practices to protect confidential information and maintain the privacy of study participants. For inquiries, please contact us at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Kanter J, Thompson AA, Pierciey FJ Jr, Hsieh M, Uchida N, Leboulch P, Schmidt M, Bonner M, Guo R, Miller A, Ribeil JA, Davidson D, Asmal M, Walters MC, Tisdale JF. Lovo-cel gene therapy for sickle cell disease: Treatment process evolution and outcomes in the initial groups of the HGB-206 study. Am J Hematol. 2023 Jan;98(1):11-22. doi: 10.1002/ajh.26741. Epub 2022 Oct 10. PMID 36161320
- [Derived] Del Pozo Martin Y. 2021 ASH annual meeting. Lancet Haematol. 2022 Feb;9(2):e92-e93. doi: 10.1016/S2352-3026(21)00384-7. Epub 2021 Dec 16. No abstract available. PMID 34922648
- [Derived] Kanter J, Walters MC, Krishnamurti L, Mapara MY, Kwiatkowski JL, Rifkin-Zenenberg S, Aygun B, Kasow KA, Pierciey FJ Jr, Bonner M, Miller A, Zhang X, Lynch J, Kim D, Ribeil JA, Asmal M, Goyal S, Thompson AA, Tisdale JF. Biologic and Clinical Efficacy of LentiGlobin for Sickle Cell Disease. N Engl J Med. 2022 Feb 17;386(7):617-628. doi: 10.1056/NEJMoa2117175. Epub 2021 Dec 12. PMID 34898139
- [Derived] Jones RJ, DeBaun MR. Leukemia after gene therapy for sickle cell disease: insertional mutagenesis, busulfan, both, or neither. Blood. 2021 Sep 16;138(11):942-947. doi: 10.1182/blood.2021011488. PMID 34115136
- [Derived] Del Pozo Martin Y. 47th Annual Meeting of the EBMT. Lancet Haematol. 2021 May;8(5):e317-e318. doi: 10.1016/S2352-3026(21)00104-6. Epub 2021 Mar 31. No abstract available. PMID 33811823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 54 participants-initiated stem cell collection and included in Intent-to-Treat (ITT) population, and of those 45 participants treated with lovo-cel and included in the transplant population.
Pre-assignment Details: Participants were enrolled as Groups A, B (B1 and B2) and C (see Reporting Groups). Since B1 and B2 contained only 2 participants and due to other factors (eg, logistical considerations), results for B1 and B2 are reported as "Group B" throughout this summary.
Groups:
- Group A: Participants who had rescue cells that were collected by bone marrow harvest method and had received treatment with lovo-cel which consists of autologous CD34+ hematopoietic stem cells (HSCs) and progenitor stem cells (PSCs) (collectively referred to as hematopoietic stem and progenitor cells or HSPCs) collected from patients with sickle cell disease (SCD) by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene (the original drug product manufacturing process for this study).
- Group B: Group B included only 2 participants treated with drug product cells collected differently and with drug product manufactured using different processes (one participant in Group B1 and one participant in Group B2 as detailed below). Note that, due to the small size of Groups B1 and B2 and due to other factors (including logistical considerations), these intermediate groups are combined as "Group B" throughout this summary for results reporting purposes.
  Group B1 participant had rescue cells and drug product cells that were collected by bone marrow harvest method and drug product was manufactured with autologous CD34+ HSPCs collected by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene. This participant's drug product was produced in 2 lots each using two different manufacturing processes (the original drug product manufacturing process and a refined drug product manufacturing process).
  Group B2 Plerixafor mobilization and apheresis were used for collection of rescue cells and exploratory manufacturing development. Participants received treatment of lovo-cel manufactured with autologous CD34+ HSPCs collected by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene (using only the refined drug product manufacturing process).
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 9 | 2 | 43
Transplant Population (TP) (TP included participants who received lovo-cel (45 TP participants).) | 7 | 2 | 36
Transplant Population for VOE (TPVOE) (TPVOE is subset of TP participants who had at least 4 protocol VOEs in the 24 months prior to Informed Consent (40 TPVOE participants).) | 6 | 2 | 32
Completed | 7 | 2 | 35
Not Completed | 2 | 0 | 8
Not completed — Withdrawal of consent | 1 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Discontinued due to failure to mobilize | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population was defined as all participants who initiate any study procedures, beginning with stem cell collection procedures (mobilization/apheresis or bone marrow harvest).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 9 | 2 | 43 | 54
Age, Continuous [Median (Full Range); unit: years] | 26.0 [18 to 43] | 24.5 [22 to 27] | 24.0 [12 to 38] | 25.0 [12 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 18 | 20
  Male | 7 | 2 | 25 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 2 | 39 | 50
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 39 | 48
  White | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Group C Participants Who Achieved Complete Resolution of Vaso-occlusive Events (VOE-CR)
Description: VOE-CR was defined as complete resolution of adjudicated VOEs between 6 months and 18 months post lovo-cel infusion. All reported VOEs were also adjudicated by an independent Event Adjudication Committee for purposes of endpoint analysis. VOEs were determined by adjudication committee after referring to protocol VOE. The committee was responsible for VOE assessment and determining whether an event met criteria for a VOE for all reported events.
Time Frame: From 6 months to 18 months post lovo-cel infusion
Population: TPVOE was subset of TP participants who had at least 4 protocol VOEs in the 24 months prior to Informed Consent.TP included participants who received lovo-cel. As per planned analysis in SAP, data was analyzed and reported for Group C participants. Analysis of efficacy endpoint for Group C was planned to be reported based on the adjudicated vaso-occlusive events (VOEs).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 32
percentage of participants | 87.5 [71.0 to 96.5]

2. Secondary Outcome: Percentage of Group C Participants With Complete Resolution of Severe VOEs (sVOE-CR)
Description: sVOE-CR was defined as the complete resolution of sVOEs, in the 6 to 18 months post lovo-cel infusion. All reported VOEs (including sVOEs) were adjudicated by an independent Event Adjudication Committee for purposes of endpoint analysis (referred to as Adjudicated sVOEs). sVOE were determined by adjudication committee after referring to protocol definition of sVOE. The committee was responsible for VOE assessment and determining whether an event met criteria for an sVOE for all reported events.
Time Frame: From 6 months to 18 months post lovo-cel infusion
Population: TPVOE was subset of TP participants who had at least 4 protocol VOEs in the 24 months prior to Informed Consent.TP included participants who received lovo-cel. As per planned analysis in SAP, data was analyzed and reported for Group C participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 32
percentage of participants | 93.8 [79.2 to 99.2]

3. Secondary Outcome: Percentage of Group C Participants Who Achieved Globin Response
Description: Globin Response is defined as meeting the following criteria for a continuous period of at least 6 months post lovo-cel infusion (starting at least 60 days after last packed red blood cell [pRBC] transfusion):
  1. Weighted average HbAT87Q percentage of non-transfused total Hb >=30% AND
  2. Weighted average non-transfused total Hb increase of >=3 g/dL compared to baseline total Hb OR weighted average non-transfused total Hb >=10 g/dL
Time Frame: From at least 60 days after last pRBC transfusion up to Month 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis, data was analyzed and reported only for TP Group C participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 36
percentage of participants | 86.1 [70.5 to 95.3]

4. Secondary Outcome: Percentage of Group C Participants Who Meet the Definition of Globin Response at Month 24
Description: Globin Response at Month 24 was defined as continuously meeting the following criteria from the first date of globin response initiating to Month 24 assessment post lovo-cel infusion:
  1. Weighted average HbAT87Q percentage of non-transfused total Hb >=30% AND
  2. Weighted average non-transfused total Hb increase of >=3 g/dL compared to baseline total Hb OR weighted average non-transfused total Hb >=10 g/dL
Time Frame: From first date of Globin Response to Month 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis, data was analyzed and reported only for TP Group C participants. Here, "Overall number of participants analyzed" signifies TP Group C participants who achieved Globin Response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 31
percentage of participants | 96.8 [83.3 to 99.9]

5. Secondary Outcome: Duration of Globin Response in Group C Participants
Description: Duration of Globin Response is the time period from the first date of Globin Response initiating to the date of last high pressure liquid chromatography (HPLC) assessment such that the weighted average HbAT87Q (%) in non-transfused total Hb and non-transfused total Hb continuously meet Globin Response criteria.
  1. Weighted average HbAT87Q percentage of non-transfused total Hb >=30% AND
  2. Weighted average non-transfused total Hb increase of >=3 g/dL compared to baseline total Hb OR weighted average non-transfused total Hb >=10 g/dL
Time Frame: From first date of Globin Response to Month 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis, data was analyzed and reported only for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who achieved Globin Response.
Measure: Median (Full Range); unit: months
Arm/Group | Group C
Number analyzed (Participants) | 31
months | 20.47 [14.7 to 23.5]

6. Secondary Outcome: Change From Baseline in the Annualized Number of VOEs in Group C Participants
Description: Change from baseline in the annualized number of VOEs was assessed from 24 months post lovo-cel infusion compared to the 24 months prior to Informed Consent. All reported VOEs were also adjudicated by an independent event adjudication committee for purposes of outcome analysis. VOEs were determined by adjudication committee after referring to protocol definition of VOE. The committee was responsible for VOE assessment and determining whether an event met criteria for a VOE for all reported events.
Time Frame: From Baseline up to 24 months post lovo-cel infusion
Population: TPVOE was subset of TP participants who had at least 4 protocol VOEs in the 24 months prior to Informed Consent.TP included participants who received lovo-cel. As per planned analysis, data was analyzed and reported for TPVOE Group C participants.
Measure: Median (Full Range); unit: Number of VOEs/year
Arm/Group | Group C
Number analyzed (Participants) | 32
Number of VOEs/year | -3.50 [-14.6 to -1.1]

7. Secondary Outcome: Change From Baseline in the Annualized Number of sVOEs in Group C Participants
Description: Change from baseline in the annualized number of sVOEs was assessed from 24 months post lovo-cel infusion compared to the 24 months prior to Informed Consent. All reported VOEs (including sVOEs) were adjudicated by an independent Event Adjudication Committee for purposes of endpoint analysis. sVOE were determined by adjudication committee after referring to protocol definition of sVOE. The committee was responsible for VOE assessment and determining whether an event met criteria for an sVOE for all reported events.
Time Frame: From Baseline up to 24 months post lovo-cel infusion
Population: as for outcome 6
Measure: Median (Full Range); unit: Number of sVOEs/year
Arm/Group | Group C
Number analyzed (Participants) | 32
Number of sVOEs/year | -3.00 [-13.0 to -0.5]

8. Secondary Outcome: Percentage of Group C Participants With Complete Resolution of VOE Between 6 and 24 Months Post Lovo-cel Infusion (VOE-CR24)
Description: VOE-CR24, defined as complete resolution of VOE between 6 months and 24 months post lovo-cel infusion. All reported VOEs were also adjudicated by an independent Event Adjudication Committee for purposes of outcome analysis. VOEs were determined by adjudication committee after referring to protocol definition of VOE. The committee was responsible for VOE assessment and determining whether an event met criteria for a VOE for all reported events.
Time Frame: From 6 months to 24 months post lovo-cel infusion
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group C:: Plerixafor mobilization and apheresis were used for collection of rescue cells, and drug product. Participants received treatment of lovo-cel manufactured with autologous CD34+ HSPCs collected by plerixafor mobilization and apheresis transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene using a further refined manufacturing process similar to commercial manufacturing.
Arm/Group | Group C:
Number analyzed (Participants) | 32
percentage of participants | 84.4 [67.2 to 94.7]

9. Secondary Outcome: Percentage of Group C Participants With Complete Resolution of sVOEs Between 6 and 24 Months Post Lovo-cel Infusion (sVOE-CR24)
Description: sVOE-CR24, defined as complete resolution of sVOEs in 6 to 24 months post lovo-cel infusion compared to the 24 months prior to Informed Consent. All reported VOEs (including sVOEs) were adjudicated by an independent Event Adjudication Committee for purposes of outcome analysis. sVOE were determined by adjudication committee after referring to protocol definition of sVOE. The committee was responsible for VOE assessment and determining whether an event met criteria for an sVOE for all reported events.
Time Frame: From 6 months to 24 months post lovo-cel infusion
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 32
percentage of participants | 90.6 [75.0 to 98.0]

10. Secondary Outcome: Percentage of Group C Participants With At Least 75% Reduction in Annualized sVOEs (sVOE-75)
Description: sVOE-75, defined as at least a 75% reduction in annualized sVOEs in the 24 months post lovo-cel infusion compared to the 24 months prior to Informed Consent. All reported VOEs (including sVOEs) were adjudicated by an independent Event Adjudication Committee for purposes of outcome analysis. sVOE were determined by adjudication committee after referring to protocol definition of sVOE. The committee was responsible for VOE assessment and determining whether an event met criteria for an sVOE for all reported events.
Time Frame: Up to 24 months post lovo-cel infusion
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 32
percentage of participants | 93.8 [79.2 to 99.2]

11. Secondary Outcome: Change From Baseline in Annualized VOE-related Hospital Admissions in Group C Participants
Description: Change from baseline was calculated as annualized number of VOE-related hospital admissions during post-drug product infusion discharge through the last study visit minus annualized number of VOE related hospital admissions at baseline. Baseline was annualized number of VOE-related hospital admissions in 24 months prior to the Informed Consent.
Time Frame: From post hospital discharge to Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: hospital admissions per year
Arm/Group | Group C
Number analyzed (Participants) | 32
hospital admissions per year | -3.00 [-13.5 to -0.5]

12. Secondary Outcome: Change From Baseline in Annualized VOE-related Total Days Hospitalized in Group C Participants
Description: Change from baseline was calculated as annualized number of VOE-related hospital days during post-drug product infusion discharge through the last study visit minus annualized number of VOE related hospital days at baseline. Baseline was annualized number of VOE-related hospital days in 24 months prior to the Informed Consent.
Time Frame: From post hospital discharge to Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: hospitalized days per year
Arm/Group | Group C
Number analyzed (Participants) | 32
hospitalized days per year | -16.75 [-136.0 to -1.5]

13. Secondary Outcome: Weighted Average of Non-transfused Total Hb in Group C Participants
Description: Non-transfused total Hb was the total g/dL of HbS + HbF + HbA2 + HbAT87Q for participants without beta + allele or HbS + HbF + HbA2 + HbAT87Q + HbA for participants with beta + allele.
Time Frame: At Month 6, 12, 18, and 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refer to the participants who were evaluable at specified time points. Evaluable participants are defined as participants who have weighted average of non-transfused total Hb at Month 6, 12, 18 and 24.
Measure: Median (Full Range); unit: gram per deciliter (g/dL)
Arm/Group | Group C
Number analyzed (Participants) | 36
gram per deciliter (g/dL)
  At Month 6 | 10.73 [5.1 to 13.1]
  At Month 12 | 11.53 [5.1 to 14.4]
  At Month 18: number analyzed (Participants) | 35
  At Month 18 | 11.70 [9.6 to 15.1]
  At Month 24: number analyzed (Participants) | 34
  At Month 24 | 11.53 [9.2 to 15.4]

14. Secondary Outcome: Weighted Average of HbS Percentage (%) in Non-transfused Total Hb in Group C Participants
Description: HbS % in non-transfused total Hb = (HbS/ non-transfused total Hb)*100.
Time Frame: At Month 6, 12, 18, and 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refer to the participants who were evaluable at specified time points. Evaluable participants are defined as participants who have weighted average of HbS % in Non-transfused Total Hb at Month 6, 12, 18 and 24.
Measure: Median (Full Range); unit: percentage of non-transfused total HbS
Arm/Group | Group C
Number analyzed (Participants) | 36
percentage of non-transfused total HbS
  At Month 6 | 50.17 [31.4 to 66.2]
  At Month 12 | 50.77 [31.4 to 68.1]
  At Month 18: number analyzed (Participants) | 35
  At Month 18 | 50.51 [39.2 to 68.1]
  At Month 24: number analyzed (Participants) | 34
  At Month 24 | 51.16 [37.8 to 61.7]

15. Secondary Outcome: Percentage of Group C Participants Who Achieved <= 70%, <= 60%, and <= 50% Weighted Average of HbS % in Non-transfused Total Hb
Description: HbS % in non-transfused total Hb = (HbS/ non-transfused total Hb)*100. The denominator of the percentage is based on the total number of participants who have non-missing value at the Visit.
Time Frame: At Month 6, 12, 18, and 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refer to the participants who were evaluable at specified time points. Evaluable participants are defined as participants who achieved <= 70%, <= 60%, and <= 50% HbS at Month 6, 12, 18 and 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Group C
Number analyzed (Participants) | 36
Percentage of participants
  At Month 6:<=70% Weighted Average HbS | 100.0
  At Month 6:<=60% Weighted Average HbS | 94.4
  At Month 6:<=50% Weighted Average HbS | 47.2
  At Month 12:<=70% Weighted Average HbS | 100
  At Month 12:<=60% Weighted Average HbS | 94.4
  At Month 12:<=50% Weighted Average HbS | 41.7
  At Month 18:<=70% Weighted Average HbS: number analyzed (Participants) | 35
  At Month 18:<=70% Weighted Average HbS | 100
  At Month 18:<=60% Weighted Average HbS: number analyzed (Participants) | 35
  At Month 18:<=60% Weighted Average HbS | 94.3
  At Month 18:<=50% Weighted Average HbS: number analyzed (Participants) | 35
  At Month 18:<=50% Weighted Average HbS | 45.7
  At Month 24:<=70% Weighted Average HbS: number analyzed (Participants) | 34
  At Month 24:<=70% Weighted Average HbS | 100
  At Month 24:<=60% Weighted Average HbS: number analyzed (Participants) | 34
  At Month 24:<=60% Weighted Average HbS | 94.1
  At Month 24:<=50% Weighted Average HbS: number analyzed (Participants) | 34
  At Month 24:<=50% Weighted Average HbS | 44.1

16. Secondary Outcome: Weighted Average of HbAT87Q % in Non-transfused Total Hb in Group C Participants
Description: HbAT87Q % in non-transfused total Hb was calculated as: HbAT87Q / non-transfused total Hb *100.
Time Frame: At Month 6, 12, 18, and 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refer to the participants who were evaluable at specified time points. Evaluable participants are defined as participants who have weighted average of HbAT87Q % in Non-transfused Total Hb at Month 6, 12, 18 and 24.
Measure: Median (Full Range); unit: percentage of non-transfused total Hb
Arm/Group | Group C
Number analyzed (Participants) | 36
percentage of non-transfused total Hb
  At Month 6 | 46.33 [25.9 to 63.0]
  At Month 12 | 46.25 [24.5 to 63.0]
  At Month 18: number analyzed (Participants) | 35
  At Month 18 | 45.99 [24.5 to 59.0]
  At Month 24: number analyzed (Participants) | 34
  At Month 24 | 45.05 [26.9 to 58.9]

17. Secondary Outcome: Weighted Average of Non-HbS % in Non-transfused Total Hb in Group C Participants
Description: Non-HbS percentage in non-transfused total Hb = [(HbF + HbA2 + HbAT87Q)/ non-transfused total Hb] *100. For participants with beta + allele, HbA was also included in the calculated for "non-HbS" for samples taken >= 60 days after last pRBC transfusion.
Time Frame: At Month 6, 12, 18, and 24 post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refer to the participants who were evaluable at specified time points. Evaluable participants are defined as participants who have weighted average of Non-HbS % in Non-transfused Total Hb at Month 6, 12, 18 and 24.
Measure: Median (Full Range); unit: percentage of non-HbS in total Hb
Arm/Group | Group C
Number analyzed (Participants) | 36
percentage of non-HbS in total Hb
  Month 6 | 49.83 [33.8 to 68.6]
  Month 12 | 49.23 [31.9 to 68.6]
  Month 18: number analyzed (Participants) | 35
  Month 18 | 49.49 [31.9 to 60.8]
  Month 24: number analyzed (Participants) | 34
  Month 24 | 48.84 [38.3 to 62.2]

18. Secondary Outcome: Non-transfused Total Hb (g/dL) Over Time
Description: as for outcome 13
Time Frame: From infusion up to Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants.
Measure: Median (Full Range); unit: g/dL
Arm/Group | Group C:
Number analyzed (Participants) | 36
g/dL | 11.80 [6.6 to 16.2]

19. Secondary Outcome: HbS % in Non-transfused Total Hb Over Time
Description: HbS (%) in non-transfused total Hb = (HbS / non-transfused total Hb)*100.
Time Frame: From infusion up to Month 24
Population: as for outcome 18
Measure: Median (Full Range); unit: Percent
Arm/Group | Group C:
Number analyzed (Participants) | 36
Percent | 51.47 [29.1 to 62.0]

20. Secondary Outcome: HbAT87Q % in Non-transfused Total Hb Over Time
Description: HbAT87Q (%) in Non-transfused total Hb = (HbAT87Q / non-transfused total Hb)*100.
Time Frame: From infusion up to Month 24
Population: as for outcome 18
Measure: Median (Full Range); unit: Percent
Arm/Group | Group C
Number analyzed (Participants) | 36
Percent | 46.01 [26.9 to 63.2]

21. Secondary Outcome: Non-HbS % of Non-transfused Total Hb Over Time
Description: Non-HbS % in non-transfused total Hb = [(HbF + HbA2 + HbAT87Q)/ non-transfused total Hb] *100.
Time Frame: From infusion up to Month 24
Population: as for outcome 18
Measure: Median (Full Range); unit: Percent
Arm/Group | Group C
Number analyzed (Participants) | 36
Percent | 48.53 [38.0 to 70.9]

22. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count in Group C Participants
Description: Reticulocytes are immature RBCs that develop in the bone marrow and circulate in the bloodstream for about a day before developing into mature RBCs. Due to the loss of mature RBCs during hemolysis, there is usually a high demand to produce new RBCs in subjects with SCD, resulting in higher than normal absolute reticulocyte counts. For this outcome Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who have absolute reticulocyte count at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: cells*10^9 per liter (cells*10^9/L)
Arm/Group | Group C
Number analyzed (Participants) | 36
cells*10^9 per liter (cells*10^9/L)
  Change at Month 12: number analyzed (Participants) | 34
  Change at Month 12 | -86.52 [-425.7 to 154.0]
  Change at Month 24: number analyzed (Participants) | 35
  Change at Month 24 | -77.95 [-344.8 to 91.0]

23. Secondary Outcome: Change From Baseline in Percent (%) Reticulocyte/Erythrocytes in Group C Participants
Description: Reticulocytes are immature RBCs that develop in the bone marrow and circulate in the bloodstream for about a day before developing into mature RBCs. The fraction of reticulocytes/erythrocytes in the blood is normally 0.5% to 2.5%, and is increased when there is peripheral hemolytic anemia. Due to the loss of mature RBCs during hemolysis, there is usually a high demand to produce new RBCs in subjects with SCD, resulting in higher than normal reticulocyte counts. For this outcome, Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who achieved % Reticulocyte/Erythrocytes at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: Percent
Arm/Group | Group C
Number analyzed (Participants) | 36
Percent
  Change at Month 12: number analyzed (Participants) | 34
  Change at Month 12 | -4.595 [-20.900 to 4.905]
  Change at Month 24: number analyzed (Participants) | 35
  Change at Month 24 | -4.847 [-18.151 to 3.077]

24. Secondary Outcome: Change From Baseline in Total Bilirubin in Group C Participants
Description: Reduction of red blood cell sickling with lovo-cel has the potential to reduce or eliminate downstream complications, including hemolysis. Total Bilirubin is a marker of RBC hemolysis and so increases in Total Bilirubin levels suggests increased hemolysis. For this outcome, Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who achieved total bilirubin count at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: milligram per deciliter (mg/dL)
Arm/Group | Group C
Number analyzed (Participants) | 36
milligram per deciliter (mg/dL)
  Change at Month 12 | -1.850 [-6.60 to 1.10]
  Change at Month 24: number analyzed (Participants) | 35
  Change at Month 24 | -1.800 [-5.80 to 0.70]

25. Secondary Outcome: Change From Baseline in Haptoglobin in Group C Participants
Description: Reduction of red blood cell sickling with lovo-cel has the potential to reduce or eliminate downstream complications, including hemolysis. Haptoglobin is a marker of RBC hemolysis and so increases in Haptoglobin levels suggests increased hemolysis. For this outcome, Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection. It should be noted that Baseline haptoglobin levels may be impacted by a range of factors that result in variability, including (but not limited to) other therapies that a participant receives (such as blood transfusions or hydroxyurea), which limit interpretability of these data.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who achieved haptoglobin count at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Group C
Number analyzed (Participants) | 36
mg/dL
  Change at Month 12: number analyzed (Participants) | 31
  Change at Month 12 | 0.0 [-26.0 to 110.0]
  Change at Month 24: number analyzed (Participants) | 32
  Change at Month 24 | 0.0 [-69.0 to 174.0]

26. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) in Group C Participants
Description: Reduction of red blood cell sickling with lovo-cel has the potential to reduce or eliminate downstream complications, including hemolysis. Lactate Dehydrogenase is a marker of RBC hemolysis and so increases in LDH levels suggests increased hemolysis, For this outcome, Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who achieved lactate dehydrogenase count at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: units per liter (U/L)
Arm/Group | Group C
Number analyzed (Participants) | 36
units per liter (U/L)
  Change at Month 12 | -147.0 [-873.0 to 102.0]
  Change at Month 24: number analyzed (Participants) | 31
  Change at Month 24 | -145.0 [-846.0 to 218.0]

27. Secondary Outcome: Change From Baseline in Cardiac T2* on MRI in Group C Participants
Description: Particulate intracellular iron causes shortening of the magnetic resonance relaxation parameter T2 due to microscopic magnetic field inhomogeneity. A myocardial T2 value of 40 msec, which equates to 0.50 mg/g of dry weight iron has widely been used as the normal mean. Myocardial T2. Values below 20 msec are considered abnormal, and values below 10 msec indicate high risk of cardiac morbidity and mortality. For this outcome, Baseline was defined as the first assessment on or after Informed Consent but before initiation of stem cell collection. If no records at screening, the last assessment prior to Informed Consent was used.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who had Cardiac T2 at Month 24.
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | Group C
Number analyzed (Participants) | 18
milliseconds (msec) | 0.00 [-18.0 to 13.0]

28. Secondary Outcome: Change From Baseline in Serum Ferritin in Group C Participants
Description: Serum ferritin is commonly used for an indirect estimation of body iron stores. Although sensitive, it is not specific for iron overload as it can be elevated in a variety of infectious and inflammatory states, and in the presence of cytolysis. For this outcome, Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who achieved serum ferritin count at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | Group C
Number analyzed (Participants) | 36
nanogram per milliliter (ng/mL)
  Change at Month 12: number analyzed (Participants) | 33
  Change at Month 12 | 1133.9 [-927.0 to 9596.0]
  Change at Month 24: number analyzed (Participants) | 34
  Change at Month 24 | 604.6 [-1328.0 to 7498.0]

29. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) by Magnetic Resonance Imaging (MRI) in Group C Participants
Description: Liver Iron Concentration of greater than 15 mg per gram dry weight (mg/g) is associated with an increased risk of hepatic disease and cardiac toxicity, whereas levels between 7 to 15 mg/g enhance the risk of hepatic fibrosis and endocrine complications. Liver Iron Concentration of greater than 1.8 mg/g dry weight is considered abnormal; however, organ damage generally does not occur with levels less than 7 mg/g. For this outcome, Baseline was defined as the first assessment on or after Informed Consent but before initiation of stem cell collection. If no records at screening, the last assessment prior to Informed Consent was used.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who achieved liver iron concentration at Month 24.
Measure: Median (Full Range); unit: milligram per gram (mg/g)
Arm/Group | Group C
Number analyzed (Participants) | 21
milligram per gram (mg/g) | 1.100 [-10.20 to 9.93]

30. Secondary Outcome: Change From Baseline in Annualized Volume of pRBC Transfusions in Group C Participants
Description: Change from baseline was calculated as annualized volume of pRBC transfusions in 6 to 24 months post lovo-cel infusion - annualized volume of pRBC transfusions at baseline. Baseline was the annualized volume of pRBC transfusion in the 24 months prior to the Informed Consent.
Time Frame: From 6 months through 24 months post lovo-cel infusion
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants with >=1 pRBC Transfusion.
Measure: Median (Full Range); unit: mL/kg/year
Arm/Group | Group C
Number analyzed (Participants) | 34
mL/kg/year | -23.60 [-522.1 to 43.3]

31. Secondary Outcome: Change From Baseline in Annualized Number of Packed Red Blood Cell (pRBC) Transfusions in Group C Participants
Description: Change from baseline was calculated as annualized number of pRBC transfusions in 6 to 24 months post lovo-cel infusion - annualized number of pRBC transfusions at baseline. Baseline was the annualized number of pRBC transfusion in the 24 months prior to the Informed Consent.
Time Frame: From 6 months through 24 months post lovo-cel infusion
Population: as for outcome 30
Measure: Median (Full Range); unit: number of pRBC transfusions/year
Arm/Group | Group C
Number analyzed (Participants) | 34
number of pRBC transfusions/year | -3.25 [-17.0 to 7.1]

32. Secondary Outcome: Change From Baseline in Erythropoietin Levels in Group C Participants
Description: Erythropoietin is a hormone produced mainly by the kidneys in response to hypoxia, which can be caused by anemia. Patients with SCD typically produce higher than normal levels of serum erythropoietin. Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who have erythropoietin levels at Baseline and at Months 12 and 24
Measure: Median (Full Range); unit: units per liter (U/L)
Arm/Group | Group C
Number analyzed (Participants) | 12
units per liter (U/L)
  Change at Month 12 | -26.20 [-286.0 to 3.0]
  Change at Month 24 | -16.55 [-276.4 to 42.0]

33. Secondary Outcome: Change From Baseline in Cardiac-pulmonary Function Via Left Ventricular Ejection Fraction (LVEF) in Group C Participants
Description: LVEF is the central measure of left ventricular systolic function. LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). This was measured by ECHO. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection. If no records at screening, the last assessment prior to Informed Consent was used.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" refers to the participants who had LVEF at Month 24
Measure: Median (Full Range); unit: percent
Arm/Group | Group C
Number analyzed (Participants) | 35
percent | -0.50 [-25.9 to 11.0]

34. Secondary Outcome: Change From Baseline in Serum Transferrin Receptor in Group C Participants
Description: Transferrin is a circulating iron carrier protein, delivering iron to cells via the transferrin receptor, and levels of serum transferrin receptor have been used as an indicator of excess iron in the body. Additionally, the transferrin receptor is highly expressed in erythroblasts, and increased levels of the soluble form (serum transferrin receptor) have been shown to be associated with increased levels of erythropoiesis. Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who had serum transferrin receptor count at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Group C
Number analyzed (Participants) | 36
milligrams per deciliter (mg/dL)
  Change at Month 12 | -0.409 [-3.35 to 0.09]
  Change at Month 24: number analyzed (Participants) | 25
  Change at Month 24 | -0.422 [-1.64 to 0.13]

35. Secondary Outcome: Change From Baseline in Renal Function as Measured by Estimated Glomerular Filtration Rate (eGFR) in Group C Participants
Description: eGFR was calculated by chronic kidney disease epidemiology collaboration (CKD-EPI) formula for participants >=18 years of age and Schwartz formula was used for participants <18 years of age. Baseline is the first assessment on or after Informed Consent but before initiation of stem cell collection. If no records at screening, the last assessment prior to Informed Consent was used.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "number analyzed" refers to the participants who had renal function at Baseline and at Months 12 and 24.
Measure: Median (Full Range); unit: milliliter/minute/1.73 square meter
Arm/Group | Group C
Number analyzed (Participants) | 36
milliliter/minute/1.73 square meter
  Change at Month 12 | -2.20 [-34.8 to 55.7]
  Change at Month 24: number analyzed (Participants) | 35
  Change at Month 24 | -7.71 [-58.7 to 43.8]

36. Secondary Outcome: Number of Participants With Shift From Baseline in Cardiac-pulmonary Function Via Echocardiogram (Tricuspid Regurgitant Jet Velocity [TRJV]) in Group C Participants
Description: TRJV over time for each participant was classified into 2 categories: <2.5 m/sec versus >=2.5 m/sec. Higher value of TRJV indicates worse result. A TRJV value of >2.5 m/s was associated with a higher risk of complications, especially in participants with Sickle Cell Disease due to hemolysis and pulmonary hypertension. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection. If no records at screening, the last assessment prior to Informed Consent was used.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" refers to the participants who had shift at baseline for TRJV at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Group C
Number analyzed (Participants) | 13
Participants
  TRJV at Baseline (<2.5 m/sec) to TRJV at Month 24 (<2.5 m/sec) | 5
  TRJV at Baseline (>=2.5 m/sec) to TRJV at Month 24 (<2.5 m/sec) | 4
  TRJV at Baseline (<2.5 m/sec) to TRJV at Month 24 (>=2.5 m/sec) | 0
  TRJV at Baseline (>=2.5 m/sec) to TRJV at Month 24 (>=2.5 m/sec) | 4

37. Secondary Outcome: Number of Participant With Shift From Baseline in Cardiac-pulmonary Function Via Pulmonary Function Tests (PFTs) in Group C Participants
Description: PFTs over time of each participant were classified into one of the five categories: normal, obstructive, restrictive, mixed obstructive and restrictive and isolated low DLco (carbon monoxide diffusing capacity). Only non-zero values are reported here. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection. If no records at screening, the last assessment prior to Informed Consent was used.
  Note: while data are provided for this outcome measure, the results for this outcome are not anticipated to be fully mature until extended participant long-term follow-up in Study LTF-307 has been achieved. The results presented below should be interpreted in that context.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" refers to the participants who had shift from baseline in PFTs at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Group C
Number analyzed (Participants) | 32
Participants
  Restrictive at Baseline to Normal at Month 24 | 2
  Restrictive at Baseline to Restrictive at Month 24 | 12
  Restrictive at Baseline to Isolated low DLco at Month 24 | 1
  Restrictive at Baseline to Not Specified at Month 24 | 3
  Isolated low DLco at Baseline to Restrictive at Month 24 | 1
  Isolated low DLco at Baseline to Isolated low DLco at Month 24 | 2
  Not Specified at Baseline to Normal at Month 24 | 2
  Not Specified at Baseline to Restrictive at Month 24 | 1
  Not Specified at Baseline to Isolated low DLco at Month 24 | 1
  Not Specified at Baseline to Not Specified at Month 24 | 7

38. Secondary Outcome: Change From Baseline in Meters Walked During 6-minute Walk Test in Group C Participants
Description: The 6-minute walk test measures the distance in meters walked during 6 minutes and can be used to assess pulmonary function. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 12 and Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome and "number analyzed" refer to the participants walked during 6-minute walk test at Baseline and at Months 12 and 24
Measure: Median (Full Range); unit: meters
Arm/Group | Group C
Number analyzed (Participants) | 25
meters
  Change at Month 12: Distance Walked in 6 Minutes | -7.13 [-62.6 to 44.4]
  Change at Month 24: Distance Walked in 6 Minutes: number analyzed (Participants) | 24
  Change at Month 24: Distance Walked in 6 Minutes | -0.65 [-46.9 to 91.0]

39. Secondary Outcome: Change From Baseline in Patient-reported Quality of Life as Measured by Patient Reported Outcomes Measurement Information System-57 (PROMIS-57): Domain (T- Score) in Group C Participants
Description: The PROMIS-57 profile was a self-reported questionnaire assessing quality of life in various 7 domains (pain interference, physical function, sleep disturbance, Ability to participate in social roles and activities, anxiety, depression, and fatigue) in participants >=18 years old.These 7 domains are scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. The higher of the T-score: the better of physical function, satisfaction with participation in social roles, and ability of participate in social roles in activities; The higher of the T-score: the worse of anxiety, depression, fatigue, sleep disturbance, and pain interference. A negative value indicates improvement, and a positive value indicates no improvement in condition. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome and "number analyzed" refer to the participants who had domain scores at Month 24.
Measure: Median (Full Range); unit: T-score
Arm/Group | Group C
Number analyzed (Participants) | 28
T-score
  Change at Month 24 (T-score): Pain Interference: number analyzed (Participants) | 27
  Change at Month 24 (T-score): Pain Interference | -7.40 [-25.5 to 13.5]
  Change at Month 24 (T-score): Physical Function: number analyzed (Participants) | 27
  Change at Month 24 (T-score): Physical Function | 5.10 [-6.5 to 17.7]
  Change at Month 24 (T-score): Sleep Disturbance: number analyzed (Participants) | 26
  Change at Month 24 (T-score): Sleep Disturbance | -4.15 [-18.8 to 16.2]
  Change at Month 24 (T-score): Ability to participate in social roles and activities: number analyzed (Participants) | 3
  Change at Month 24 (T-score): Ability to participate in social roles and activities | 10.60 [7.8 to 20.9]
  Change at Month 24 (T-score): Anxiety: number analyzed (Participants) | 27
  Change at Month 24 (T-score): Anxiety | 0.00 [-24.3 to 20.4]
  Change at Month 24 (T-score): Depression | 0.00 [-20.3 to 17.4]
  Change at Month 24 (T-score): Fatigue: number analyzed (Participants) | 27
  Change at Month 24 (T-score): Fatigue | -7.70 [-30.2 to 8.5]

40. Secondary Outcome: Change From Baseline in Patient-reported Quality of Life as Measured by PROMIS-57: Pain Intensity Score in Group C Participants
Description: The PROMIS-57 profile was a self-reported questionnaire assessing quality of life in various domains in participants >=18 years old. Pain intensity was scored from 0 to 10, with higher scores indicating greater pain intensity. A negative value indicates improvement in pain intensity and a positive value indicates no improvement or worsening in pain intensity. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome and "number analyzed" refer to the participants who had pain intensity score at Month 24.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Group C
Number analyzed (Participants) | 26
Score on a scale | -2.0 [-6 to 4]

41. Secondary Outcome: Change From Baseline in Patient-reported Quality of Life as Measured by Patient Reported Outcomes Measurement Information System- 49 (PROMIS-49)): Domain (T- Score) in Group C Participants
Description: The PROMIS-49 profile was a self-reported questionnaire assessing quality of life in various 6 domains (physical function mobility, peer relationships, pain interference, anxiety, depression, and fatigue) in participants <=18 years old. These 6 domains are scored on a 5-point Likert scale and converted into standardized T-scores with a mean of 50 and a standard deviation of 10 based on a US general population. The higher of the T-score, the better of physical function mobility, and peer relationships; The higher of the T-score, the worse of anxiety, depression symptoms, fatigue, and pain interference. A negative value indicates improvement, and a positive value indicates no improvement in condition. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who had domain scores at Month 24.
Measure: Median (Full Range); unit: T-score
Arm/Group | Group C
Number analyzed (Participants) | 4
T-score
  Change at Month 24 (T-score): Physical Function Mobility | 7.15 [-10.1 to 13.0]
  Change at Month 24 (T-score): Anxiety | -0.40 [-9.1 to 9.4]
  Change at Month 24 (T-score): Depressive Symptoms | 0.95 [-5.1 to 8.5]
  Change at Month 24 (T-score): Fatigue | -5.70 [-24.5 to 0.0]
  Change at Month 24 (T-score): Peer Relationships | 2.45 [-2.2 to 10.6]
  Change at Month 24 (T-score): Pain Interference | -2.95 [-13.6 to 2.9]

42. Secondary Outcome: Change From Baseline in Patient-reported Quality of Life as Measured by PROMIS-49: Pain Intensity Score in Group C Participants
Description: The PROMIS-49 profile was a self-reported questionnaire assessing quality of life in various domains in participants <=18 years old. Pain intensity was scored from 0 to 10, with higher scores indicating greater pain intensity. A negative value indicates improvement in pain intensity and a positive value indicates no improvement or worsening in pain intensity. Baseline was the first assessment on or after Informed Consent but before initiation of stem cell collection.
Time Frame: Baseline, Month 24
Population: TP included participants who received lovo-cel. As per planned analysis data was analyzed and reported for TP Group C participants. Here, "Overall number of participants analyzed" signifies participants who had pain intensity scores at Month 24.
Measure: Median (Full Range); unit: Score on a Scale
Arm/Group | Group C
Number analyzed (Participants) | 4
Score on a Scale | -4.0 [-7 to 0]

ADVERSE EVENTS:
Time Frame: From date of Informed Consent signing up to Month 24
Description: ITT population was defined as all participants who initiate any study procedures, beginning with stem cell collection procedures (mobilization/apheresis or bone marrow harvest).
Groups:
- Group A: Participants who had rescue cells that were collected by bone marrow harvest method and had received treatment with lovo-cel which consists of autologous CD34+ HSCs and PSCs (collectively referred to as hematopoietic stem and progenitor cells or HSPCs) collected from participants with SCD by bone marrow harvest transduced with BB305 lentiviral vector encoding the human beta-A-T87Q globin gene (the original drug product manufacturing process for this study).
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/2 | 1/43
Serious Adverse Events (participants affected / at risk) | 9/9 | 2/2 | 33/43
Other Adverse Events (participants affected / at risk) | 9/9 | 2/2 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=9) | Group B (N=2) | Group C (N=43)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 6 | 2 | 21
Long QT syndrome (Cardiac disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2
Bacteraemia (Infections and infestations) | 2 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 2
Influenza (Infections and infestations) | 1 | 0 | 3
Lung abscess (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Drug dependence (Psychiatric disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Face oedema (General disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 5
Device related thrombosis (General disorders) | 0 | 0 | 2
Drug withdrawal syndrome (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Infective thrombosis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Sedation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Psychogenic seizure (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2
Affective disorder (Psychiatric disorders) | 0 | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Catheter bacteraemia (Infections and infestations) | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=9) | Group B (N=2) | Group C (N=43)
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | 21
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 25
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 16
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 26
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 6 | 1 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 2 | 33
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 3
Vision blurred (Eye disorders) | 1 | 0 | 5
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 15
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 5
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 22
Dental caries (Gastrointestinal disorders) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 19
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 4
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 2 | 36
Oral pain (Gastrointestinal disorders) | 2 | 0 | 5
Stomatitis (Gastrointestinal disorders) | 7 | 2 | 32
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0 | 26
Catheter site pain (General disorders) | 1 | 0 | 12
Chills (General disorders) | 1 | 0 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 1 | 16
Influenza like illness (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 6
Puncture site oedema (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 1 | 20
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 3 | 0 | 3
Gastroenteritis (Infections and infestations) | 1 | 0 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 8
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 9 | 2 | 10
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 4
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1 | 3
Alanine aminotransferase increased (Investigations) | 2 | 1 | 21
Antiphospholipid antibodies positive (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 21
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 10
Blood bilirubin increased (Investigations) | 2 | 1 | 16
Blood magnesium decreased (Investigations) | 1 | 0 | 0
Blood oestrogen decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 5
Troponin T increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 14
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 7
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 14
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 19
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 3
Device issue (Product Issues) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 14
Insomnia (Psychiatric disorders) | 3 | 0 | 14
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Hydrosalpinx (Reproductive system and breast disorders) | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 16
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 10
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 15
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 5
Post procedural drainage (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 8
Hypotension (Vascular disorders) | 1 | 0 | 3
Superficial vein prominence (Vascular disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 7
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 11
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0
Skin candida (Infections and infestations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 11
Weight decreased (Investigations) | 0 | 1 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 19
Embolism (Vascular disorders) | 0 | 1 | 3
Hot flush (Vascular disorders) | 0 | 1 | 4
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 5
Palpitations (Cardiac disorders) | 0 | 0 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 6
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 5
Pain (General disorders) | 0 | 0 | 13
Peripheral swelling (General disorders) | 0 | 0 | 4
Chest pain (General disorders) | 0 | 0 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 5
Influenza (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 7
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 3
Blood follicle stimulating hormone increased (Investigations) | 0 | 0 | 3
International normalised ratio increased (Investigations) | 0 | 0 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 7
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 12
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 10
Depression (Psychiatric disorders) | 0 | 0 | 6
Panic attack (Psychiatric disorders) | 0 | 0 | 4
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02140554/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT02140554/SAP_001.pdf